CLINICAL TRIAL: NCT00205647
Title: A Phase II Multicenter Efficacy, Safety and Dose-Effect Study of the Expectorant Activity of Oral N-acetylcystein (NAC) in Patients With Stable, Chronic Bronchitis
Brief Title: Study of Expectorant Activity of Oral N-acetylcystein (NAC) in Patients With Stable Chronic Bronchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Zambon SpA (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZAM-13343
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2000-03

CONDITIONS: Chronic Bronchitis
Keywords: Chronic Bronchitis; N-acetylcysteine (NAC); Quality of Life; Mucus
MeSH Terms: conditions — Bronchitis, Chronic

INTERVENTIONS:
Drug: Oral N-acetycystein (NAC)

SUMMARY:
This is a randonmized, masked, placebo-controlled parallel group, clinical trial to evaluate the effects of three different doses of N-acetyl L-cysteine (NAC) and placebo on patient safety and on physical and transport properties of expectorated sputum. Patient sumptoms, quality of life and exacerbation will also be followed as well as pulmonary function testing and functional exercise capacity. We hypothesized that a prolongeed course of oral NAC favorably affects the morbidity of chronic bronchitis, particularly the incidence of acute exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Smokers (past or current,20 pack years) with diagnosis of chronic bronchitis
* expectorate sputum daily
* FEV1 of 40-70%
* understand and fill out questionnaire daily

Exclusion Criteria:

* other investigational within 30 days
* change in smoking habit within 6 months
* pulmonary diagnosis other that chronic bronchitis
* significant renal, cardiac, hepatic or endocrine diseases
* psychiatric disorder or evidence of alcoholism or drug abuse within year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 1997-01; Study Completion 2000-03

PRIMARY OUTCOMES:
Acute exacerbations
Clinical assessments

SECONDARY OUTCOMES:
Functional exercise capacity
Relationship between mucus physical and transport properties

CONTACTS AND LOCATIONS:
Overall Officials: Bruce K Rubin, MEng,MD,MBA, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States